CLINICAL TRIAL: NCT02802722
Title: A Prospective Randomised Placebo-controlled Study of the Influence of Vitamin D Supplementation on Resolution of Inflammation Following Community-acquired Pneumonia
Brief Title: Does Vitamin D Supplementation Enhance Resolution of Inflammation After Community-acquired Pneumonia?
Acronym: ResolveD-CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 011280
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pneumonia
Keywords: convalescence; inflammation; resolution; vitamin D
MeSH Terms: conditions — Pneumonia; Convalescence; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate supplementation (Active Comparator): Dietary supplement: Vitamin D3 supplementation - oral capsules 6400 International Units once daily for 6 weeks Peripheral blood and induced sputum sampling Chest computerised tomography (CT) scans Symptom questionnaire
  Interventions: Dietary Supplement: Vitamin D3 supplementation; Biological: Peripheral blood and induced sputum sampling; Radiation: Chest computerised tomography (CT) scans; Other: Symptom questionnaire
- Delayed supplementation (Placebo Comparator): Placebo: oral placebo capsules once daily for 6 weeks Peripheral blood and induced sputum sampling Chest computerised tomography (CT) scans Symptom questionnaire
  Interventions: Biological: Peripheral blood and induced sputum sampling; Radiation: Chest computerised tomography (CT) scans; Other: Symptom questionnaire; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 supplementation — Capsules to be dispensed using an electronic dispenser to allow real time logging of adherence.
  Other Names: cholecalciferol; colecalciferol
  Arms: Immediate supplementation
Biological: Peripheral blood and induced sputum sampling — To attain samples for immunological testing
Radiation: Chest computerised tomography (CT) scans — For volumetric quantification of lung abnormalities
Other: Symptom questionnaire — Symptom questionnaire for recent symptom history
Other: Placebo — To be dispensed using an electronic dispenser to allow real time logging of adherence.
  Arms: Delayed supplementation

SUMMARY:
Previous research has shown that people who have been hospitalised for pneumonia are more likely to die of conditions such as heart attacks, stroke and cancer in the weeks to months after their illness. This risk is linked to raised levels of inflammation. Laboratory research shows that vitamin D can help to clear inflammation. Vitamin D deficiency is very common in the United Kingdom. The investigators are conducting this study to find out if taking vitamin D can hasten long-term recovery from pneumonia by reducing inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥50 years of age
2. Vitamin D deficiency at entry, defined as a serum total 25(OH)D concentration <50 nmol/L
3. Admission to hospital with an acute illness (≤21 days) consistent with community-acquired pneumonia - at least one symptom of a lower respiratory tract infection (cough, sputum production, dyspnoea, wheeze, chest discomfort or pain, fever) and new infiltrate on chest radiograph
4. Adequate mental capacity to give informed consent for participation in the study and gives written informed consent

Exclusion Criteria:

1. Currently taking any vitamin D supplementation
2. Known HIV infection, other condition causing immunosuppression, current immunosuppressive therapy or systemic corticosteroids
3. Known malignancy not in remission for >3 years or terminal illness with prognosis <1year
4. History of smoking within the previous 1 year
5. Known or suspected diagnosis of chronic obstructive pulmonary disease (COPD)
6. Previous hospitalisation within 10 days of admission
7. Aspiration pneumonia diagnosed by the clinical team
8. Known diagnosis of cystic fibrosis, bronchiectasis or interstitial lung disease at screening
9. Complications of pneumonia such as empyema or lung abscess at entry
10. Recent acute coronary syndrome within the previous 1 month
11. Long term oxygen therapy, chronic mechanical ventilation dependency or other contraindication to sputum induction
12. Serum corrected calcium concentration >2.65 mmol/L at entry
13. Chronic kidney disease stage 4-5 (estimated glomerular filtration rate <30ml/min) on an existing blood sample from the current hospital admission
14. Known clinical diagnosis of liver failure
15. Known or suspected diagnosis of active pulmonary tuberculosis
16. Known diagnosis of primary hyperparathyroidism
17. Known diagnosis of sarcoidosis
18. Known diagnosis of nephrolithiasis
19. Taking carbamazepine, phenytoin, phenobarbital, primidone, cardiac glycosides or benzothiadiazines with concomitant calcium supplementation at entry
20. Known allergy to vitamin D or its excipients
21. Currently taking part in another research study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma IL-6 concentrations | after 6 weeks of vitamin D3 supplementation
  IL-6

SECONDARY OUTCOMES:
Serum CRP | after 6 weeks of vitamin D3 supplementation
  CRP
Total white cell count and differential white cell count in induced sputum samples | after 6 weeks of vitamin D3 supplementation
  WBC and differential counts
Immune cell phenotypes in peripheral blood | after 6 weeks of vitamin D3 supplementation
  flow cytometry phenotypes, blood
Immune cell phenotypes in induced sputum samples | after 6 weeks of vitamin D3 supplementation
  flow cytometry phenotypes, induced sputum
Plasma concentrations of pro- and anti-inflammatory mediators in peripheral blood | after 6 weeks of vitamin D3 supplementation
  Cytokines, lipid mediators, blood
Plasma concentrations of pro- and anti-inflammatory mediators in induced sputum samples | after 6 weeks of vitamin D3 supplementation
  Cytokines, lipid mediators, induced sputum
Plasma concentrations of pro- and anti-inflammatory mediators in supernatants from whole blood stimulated with antigens ex-vivo | after 6 weeks of vitamin D3 supplementation
  Cytokines, lipid mediators, stimulated blood
Whole blood transcriptional profiles | after 6 weeks of vitamin D3 supplementation
  mRNA
Volumes of lung abnormalities on chest CT imaging | after 6 weeks of vitamin D3 supplementation
  CT data
Pneumonia symptom scores | after 6 weeks of vitamin D3 supplementation
  CAP-Sym scores

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Martineau, MBBS, Study Chair — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yende S, D'Angelo G, Kellum JA, Weissfeld L, Fine J, Welch RD, Kong L, Carter M, Angus DC; GenIMS Investigators. Inflammatory markers at hospital discharge predict subsequent mortality after pneumonia and sepsis. Am J Respir Crit Care Med. 2008 Jun 1;177(11):1242-7. doi: 10.1164/rccm.200712-1777OC. Epub 2008 Mar 27. PMID 18369199
- [Background] Remmelts HH, van de Garde EM, Meijvis SC, Peelen EL, Damoiseaux JG, Grutters JC, Biesma DH, Bos WJ, Rijkers GT. Addition of vitamin D status to prognostic scores improves the prediction of outcome in community-acquired pneumonia. Clin Infect Dis. 2012 Dec;55(11):1488-94. doi: 10.1093/cid/cis751. Epub 2012 Aug 31. PMID 22942205